CLINICAL TRIAL: NCT03319342
Title: Kindness to Others or to Oneself: A Pilot Randomized Controlled Trial of Kindness Interventions to Enhance Well-Being in Breast Cancer Survivors
Brief Title: Kindness Interventions in Enhancing Well-Being in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-000560; NCI-2017-01469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID776; 17-000560 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2017-09-28; First posted 2017-10-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2019-12

CONDITIONS: Cancer Survivor; Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I (acts of kindness to others) (Experimental): Participants perform small acts of kindness or generosity for others 3 times per week for 4 weeks and complete weekly online questionnaires.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration
- Group II (acts of kindness to self) (Experimental): Participants perform small acts of kindness for themselves 3 times per week for 4 weeks and complete weekly online questionnaires.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration
- Group III (self-kindness meditation) (Experimental): Participants direct kind, loving thoughts to themselves, via guided meditation, 3 times per week for 4 weeks and complete weekly online questionnaires.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration
- Group IV (track daily activities) (Active Comparator): Participants keep track of their daily activities, focusing on factual information rather than thoughts and feelings, on 3 separate days each week. At the end of the week, participants report on their activities and complete several online questionnaires.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Perform acts of kindness to others
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group I (acts of kindness to others)
Behavioral: Behavioral Intervention — Perform acts of kindness to self
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group II (acts of kindness to self)
Behavioral: Behavioral Intervention — Perform self-kindness meditation
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group III (self-kindness meditation)
Behavioral: Behavioral Intervention — Keep track of daily activities
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group IV (track daily activities)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
Emerging evidence suggests that both extending kindness towards others and self-kindness practices may have beneficial effects on well-being. This randomized pilot clinical trial will investigate the efficacy of two kindness interventions -acts of kindness (to self or to other) and loving-kindness meditation- for use with early-stage breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To refine two interventions - loving kindness and acts of kindness- for use with breast cancer survivors using an online platform.

II. To determine the feasibility and preliminary efficacy of these interventions on positive affect, depressive symptoms, and other aspects of well-being among women with breast cancer.

OUTLINE: Participants are randomized to 1 of 4 groups.

GROUP I (ACTS OF KINDNESS TO OTHERS): Participants perform small acts of kindness or generosity for others 3 times per week for 4 weeks and complete weekly online questionnaires.

GROUP II (ACTS OF KINDNESS TO SELF): Participants perform small acts of kindness for themselves 3 times per week for 4 weeks and complete weekly online questionnaires.

GROUP III (SELF-KINDNESS MEDITATION): Participants direct kind, loving thoughts to themselves, via guided meditation, 3 times per week for 4 weeks and complete weekly online questionnaires.

GROUP IV (CONTROL): Participants keep track of their daily activities, focusing on factual information rather than thoughts and feelings, on 3 separate days each week. At the end of the week, participants report on their activities and complete several online questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women previously diagnosed with stage 0-IIIA breast cancer
* Have completed treatment with surgery, radiation, and/or chemotherapy
* Have not had a cancer recurrence
* Have access to the internet and an active email account

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (Center for Epidemiologic Studies Depression Scale) | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Depressive symptoms will be measured at baseline and post-intervention using the 20-item Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a measure of symptom severity across the previous week, and total scores range from 0 to 60. Higher scores indicate greater severity of depressive symptoms.
Psychological well-being measured by the Mental Health Continuum-Short Form | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Psychological well-being measured by the Mental Health Continuum-Short Form (MHC-SF) Well-being will be measured at both baseline and post-intervention via the 14-item MHC-SF. Total scores range from 0 to 70, with higher scores indicating greater overall well-being. The MHC-SF is comprised of three empirically derived subscales: the 3-item Emotional Well-Being Subscale (score range: 0 to 15), the 6-item Psychological Well-Being Subscale (score range: 0 to 30), and the 5-item Social Well-Being Subscale (score range: 0 to 25). Higher scores on each subscale indicate greater well-being within that domain.

SECONDARY OUTCOMES:
Big-5 Personality Dimensions measured by the Ten-Item Personality Inventory (TIPI) | Baseline
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Big-5 Personality Dimensions measured by the Ten-Item Personality Inventory (TIPI) measured at baseline: Personality dimensions will be measured at baseline by the 10-item TIPI. There are 5 subscales on the TIPI, each with 2-items: Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness to Experience. Scores on each subscale range from 2 to 14, with higher scores indicating greater endorsement of the corresponding personality domain.
Empathy measured by the Perspective Taking & Empathic Concern Subscales of the Interpersonal Reactivity Index | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Empathy measured by the Perspective Taking & Empathic Concern Subscales of the Interpersonal Reactivity Index: Empathy will be measured pre- and post-intervention using the 6-item Perspective Taking (range: 0 to 30) and 7-item Empathic Concern Subscales (range: 0-35) of the IRI. Higher scores indicate greater characteristics of empathy.
Fatigue measured by the Severity items of the Fatigue Symptom Inventory | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Fatigue measured by the Severity items of the Fatigue Symptom Inventory (FSI): Fatigue will be measured pre- and post-intervention using the 4-item Severity subscale of the FSI. Scores range from 0 to 40, with higher scores indicating greater severity.
Fulfillment of psychological needs measured by the Balanced Measure of Psychological Needs | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Fulfillment of psychological needs measured by the Balanced Measure of Psychological Needs: Fulfillment of psychological needs will be measured weekly using the 9-item Balanced Measure of Psychological Needs. Scores range from 5 to 45, with higher scores indicating greater life satisfaction.
Life satisfaction measured by the Satisfaction with Life Scale | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Life Satisfaction measured by the Satisfaction with Life Scale: Satisfaction with life will be measured pre- and post-intervention using the 5-item Satisfaction With Life Scale. Scores range from 5 to 35, with higher scores indicating greater satisfaction. A score of 31 to 35 represents "extremely satisfied," for example.
Pain measured by the Pain Subscale of the Rand Health 36-item Short Form Survey | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Pain measured by the Pain Subscale of the Rand Health 36-item Short Form Survey (SF-36): Pain severity and interference will be measured pre- and post-intervention using the 2-item pain subscale of the SF-36. Scores range from 0 to 100, with higher scores indicating less severity/interference.
Positive and negative affect measured by the Affect-Adjective Scale | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Positive and negative affect measured by the Affect-Adjective Scale: Positive and negative affect will be measured weekly using the 9-item Affect-Adjective Scale. Three additional adjectives (i.e., embarrassed, uncomfortable, ashamed) were added by the researchers. Scores on the 4-item positive affect subscale range from 0 to 24, with higher scores indicating more positive affect. Scores on the 5-item negative affect subscale range from 0 to 30, with higher scores indicating greater negative affect.
Qualitative assessment of acts performed | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Qualitative assessment of acts performed: At the end of each week, participants will be asked to report on their weekly activities via a free response text box. The content of these activities may be coded or analyzed to provide context to quantitative data.
Self-kindness measured by the Self-Compassion Scale | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Self-kindness measured by the Self-Compassion Scale (SCS): Dispositional self-kindness will be measured pre- and post-intervention using the 5-item Self-Kindness Subscale of the SCS. Total scores on the Self-Kindness Subscale range from 5 to 25, with higher scores indicating greater levels of self-compassion.
Sleep disturbance measured by the Patient-Reported Outcomes Measurement Information System Sleep Disturbance Scale | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Sleep disturbance measured by the PROMIS Sleep Disturbance Scale: Sleep disturbance will be measured pre- and post-intervention using the 4-item PROMIS Sleep Disturbance Scale. Scores range from 4 to 20, with higher scores indicating more disturbance.
Social connection measured by the Attachment Subscale of the Social Provisions Scale | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Social connection measured by the Attachment Subscale of the Social Provisions Scale: Social connection will be measured pre- and post-intervention using the 4-item Attachment subscale of the Social Provisions Scale. Scores range from 4 to 16, with higher scores indicating greater social connection.
Social support measured by the 2-way Social Support Scale | Up to 2 years
  Analyses will be conducted under the intent-to-treat principle, including all participants in their assigned condition, accomplished by fitting models to all available data for each outcome measure, including data of participants with incomplete follow-up. Linear mixed models provide valid inferences under a missing at random assumption. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. Analyses will control for any participant characteristics with baseline imbalance among conditions or that differ between participants retained.
  Social support measured by the 2-way Social Support Scale: Social support will be measured pre- and post-intervention using the 21-item 2-way Social Support Scale. Total scores range from 0 to 105, with higher scores indicating more perceived support.

CONTACTS AND LOCATIONS:
Overall Officials: Julienne Bower, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California-Riverside, Riverside, California